CLINICAL TRIAL: NCT01617551
Title: Effect of Renal Denervation on NO-mediated Regulation of Salt- and Water Excretion, Vasoactive Hormones and Tubular Transport Proteins in Patients With Resistant Hypertension
Brief Title: Effect of Renal Denervation on NO-mediated Sodium Excretion and Plasma Levels of Vasoactive Hormones
Acronym: RENO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Regional Hospital Holstebro (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, Professor, MD, Dr.Sci., Regional Hospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RENO_01
Record Dates: First submitted 2012-06-06; First posted 2012-06-12 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Essential Hypertension
Keywords: Essential hypertension; Nitric oxide; Renal denervation; Sodium; GFR
MeSH Terms: conditions — Essential Hypertension | interventions — omega-N-Methylarginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Renal denervation (Experimental): Patient group randomized to renal denervation
  Interventions: Drug: NG-monomethyl-L-arginine (L-NMMA)
- Sham (Sham Comparator): Patients randomized to sham procedure
  Interventions: Drug: NG-monomethyl-L-arginine (L-NMMA)

INTERVENTIONS:
Drug: NG-monomethyl-L-arginine (L-NMMA) — Acute L-NMMA treatment (4,5 mg/kg loading dose followed by 3 mg/kg sustain infusion for 1 hour)

SUMMARY:
Catheter based renal denervation (CRD) in humans represents a promising new treatment of resistant hypertension. CRD is currently investigated as a treatment option in patients with resistant hypertension defined as at least 3 antihypertensive drugs (including a diuretic) in a randomized, sham-controlled, multicenter trial in Denmark (ReSet). In ReSet, patients are randomized to either CRD or a sham procedure with 6 months follow up. The mechanisms by which CRD reduce blood pressure are only partly understood and the interaction between renal sympathetic nerves and nitric oxide (NO) has not been investigated in humans.

To Study the interaction between NO and renal sympathetic nerves, we designed the present substudy, where the effects of NO-inhibition on renal, hemodynamic and hormonal variables are studied before and after CRD.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-70 years
* Stable antihypertensive treatment for 1-month with at least 3 antihypertensive drugs including a diuretic
* Day-time ambulatory blood pressure > 145/75 mmHg

Exclusion Criteria:

* Non compliance
* Pregnancy/no-anticonception in fertile women
* Radiocontrast allergy
* Malignancy
* Congestive heart failure (EF < 50)
* eGFR < 45
* Unstable angina pectoris
* Recent myocardial infarction or PCI (< 6 mdr)
* Secondary hypertension
* Renal artery stenosis or multiple renal arteries on CT
* Claudication

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-03; Primary Completion 2014-03 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Fractional excretion of sodium after acute L-NMMA treatment | 1 month before and after CRD

SECONDARY OUTCOMES:
Glomerular filtration rate (GFR) before and after L-NMMA treatment | 1 month before and after CRD

CONTACTS AND LOCATIONS:
Overall Officials: Jesper N Bech, MD, Ph.D, Principal Investigator — Dept. of medical research
Locations (1):
- Dept. of medical research, Holstebro, Denmark